CLINICAL TRIAL: NCT07008872
Title: Clinical Study on the Efficacy and Safety of CD7 CAR-T Cell Therapy Targeting CD7-positive Relapsed/Refractory T Cell Lymphoma/Acute Leukemia
Brief Title: CD7 CAR-T Cell Therapy Targeting CD7-positive Relapsed/Refractory T Cell Lymphoma/Acute Leukemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qi deng (Other)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Qi deng, Chief Physician, Tianjin First Central Hospital
Organization: Tianjin First Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XB-20240912-1
Record Dates: First submitted 2025-05-19; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: CD7+ Lymphoma; CD7+ Acute Leukemia
Keywords: CD7 CART, AL, lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD7 CAR-T (Experimental): For intravenous infusion
  Interventions: Biological: CD7 CART

INTERVENTIONS:
Biological: CD7 CART — For intravenous infusion

SUMMARY:
CD7 molecules are thought to be associated with disease aggressiveness, drug resistance, and poor prognosis. Intensive chemotherapy, immunotherapy, hematopoietic stem cell transplantation (HSCT) and other treatment regimens have achieved remarkable results in the treatment of hematologic malignant diseases. Nevertheless, patients with hematologic malignancies may still tolerate acquired therapy during the above treatments, and molecular targeted immunotherapy provides a safe, efficient and specific treatment for such patients The scheme has attracted more and more researchers' attention. The use of CD7 molecules as a new target for molecularly targeted anti-tumor therapy may provide a new research direction for the treatment of CD7 relapsed/refractory hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled:

1. Subjects diagnosed with relapsed/refractory lymphoma/leukemia:

   1. Relapsed/refractory T-cell malignant lymphoma: patients who have not remission and recurrence after at least 2 courses of standardized second-line or above treatment (including hematopoietic stem cell transplantation).
   2. Relapsed/refractory T-cell acute lymphocytic or myeloid leukemia meeting any of the following criteria:

   i) Relapse: After achieving complete remission with a standard treatment regimen (including hematopoietic stem cell transplantation), blasts appear in peripheral blood or bone marrow (proportion>5%), or extramedullary diseases occur; ii) Refractory: No complete remission after at least two courses of standard induction therapy.
2. Bone marrow flow cytometry detected tumor cells as CD7 and/or extramedullary lesions with a clear diagnosis of CD7 by pathological immunohistochemistry at the time of enrollment screening;
3. If tumor cells are detected in peripheral blood during enrollment screening, flow cytometry must be used to detect that the immunophenotype of tumor cells on the surface of tumor cells is both negative for CD4 and CD8. If the immunophenotype on the surface of peripheral blood tumor cells is not CD4 and CD8 negative, the proportion of peripheral blood tumor cells must be ≤1%;
4. Expected survival greater than 3 months from the date of signing the informed consent form;
5. Subjects with a performance status of 0~2 in the Eastern Cooperative Oncology Group (ECOG) score;
6. 14 years old≤ age ≤ 75 years old, male or female;
7. HGB at least ≥70g/L, blood transfusion is available;
8. Liver and kidney function, heart and lung function meet the following requirements:

   1. creatinine ≤1.5×ULN;
   2. left ventricular ejection fraction ≥50%;
   3. Oxygen saturation >90%;
   4. Total bilirubin ≤1.5×ULN; ALT and AST ≤2.5×ULN;
9. Subject or guardian understands and signs the informed consent form.

Exclusion Criteria:

1. One of the following cardiac criteria occurs: atrial fibrillation; Myocardial infarction within the past 12 months; Prolonged QT syndrome or secondary QT Extension, to be determined by the researcher. Echocardiography with LVSF<30% or LVEF<50%; Clinically significant pericardial effusion; Heart function Incomplete NYHA III or IV (confirmed by echocardiography within 12 months after treatment);
2. Active GVHD;
3. Have a history of severe pulmonary dysfunction;
4. Merge other advanced malignant tumors;
5. Combination of severe or persistent infections that cannot be effectively controlled;
6. Combination of severe autoimmune diseases or congenital immunodeficiency;
7. Active hepatitis (hepatitis B virus deoxyribonucleic acid [HBV-DNA ≥ 500 IU/ml and abnormal liver function] or anti hepatitis C virus Positive for HCV Ab, HCV-RNA above the detection limit of the analytical method, and abnormal liver function;
8. Human immunodeficiency virus (HIV) infection or syphilis infection;
9. Have a history of severe allergies to biological products (including antibiotics);
10. There are central nervous system disorders, such as uncontrolled epilepsy, cerebral ischemia/hemorrhage, dementia, cerebellar diseases, etc;
11. Female patients who are pregnant or breastfeeding, or have a pregnancy plan within 12 months;
12. The researcher believes that there may be situations that increase the risk to the subjects or interfere with the test results.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of CD7 CAR-T cell therapy in relapsed/refractory malignant lymphoma/acute leukemia | up to one month after the CAR-T infusion
  the incidence and severity of immune therapy related toxic reactions (irAEs)
Evaluate the effcacy of CD7 CAR-T cell therapy in relapsed/refractory malignant lymphoma/acute leukemia | one month and three month after the CAR-T infusion
  CR rate on M1 and M3
Evaluate the effcacy of CD7 CAR-T cell therapy in relapsed/refractory malignant lymphoma/acute leukemia | one month and three month after the CAR-T infusion
  ORR(CR and PR) on M1 and M3

SECONDARY OUTCOMES:
long-term efficacy | up to one year after the CAR-T infusion
  DOR
long-term efficacy | up to one year after the CAR-T infusion
  PFS
long-term efficacy | up to one year after the CAR-T infusion
  OS
Cell pharmacokinetics Dynamic indicators | Day7, Day10, Day14, Day28 after the CAR-T infusion
  CAR-T/T% by flow cytometry
Cell pharmacokinetics Dynamic indicators | Day7, Day10, Day14, Day28 after the CAR-T infusion
  CARgene copy numbers by qPCR
Cell pharmacokinetics Dynamic indicators | up to one month after the CAR-T infusion
  Area under the plasma concentration versus time curve(AUC)
Cell pharmacokinetics Dynamic indicators | up to one mpnth after the CAR-T infusion
  Peak Plasma Concentration (Cmax)